CLINICAL TRIAL: NCT06887335
Title: An Observational Prospective Study on the Safety and Feasibility of Deep Sedation Under Proceduralist Direction With Pre-emptive Endotracheal Intubation for Advanced Bronchoscopy Procedures
Brief Title: Deep Sedation With Pre-emptive Endotracheal Intubation for Advanced Bronchoscopy Procedures
Status: Recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Hee Yun Seol, Assistant professor for fund, Pusan National University Yangsan Hospital
Other Study IDs: 11-2025-013
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring a bronchoscopy-assisted procedure for diagnostic or therapeutic purposes
  Interventions: Procedure: Deep Sedation Under Proceduralist Direction with Pre-emptive Endotracheal Intubation

INTERVENTIONS:
Procedure: Deep Sedation Under Proceduralist Direction with Pre-emptive Endotracheal Intubation — If an eligible subject consents to participate in the study, deep sedation and preemptive endotracheal intubation will be performed, followed by bronchoscopy. Deep sedation will be administered according to the study protocol, with final approval of sedative administration given by the proceduralist. Oxygen will be supplied at a flow rate of 4-6 L/min via a nasal cannula before sedative administration.
  To achieve a deep sedation state (Modified Observer's Assessment of Alertness/Sedation [MOAA/S] score ≤ 2, defined as the patient not opening their eyes despite repeated verbal stimuli), an initial dose of 50 mcg fentanyl will be administered, followed by 2.5-5 mg of remimazolam. The sedation depth will be assessed every two minutes using the MOAA/S score. If the patient has not reached deep sedation, an additional 2.5 mg of remimazolam will be administered.
  Once deep sedation is achieved, lidocaine will be sprayed onto the trachea and bronchi using a bronchoscope for local anesthe

SUMMARY:
Bronchoscopy is crucial for diagnosing and treating respiratory diseases and is recommended under sedation. Deep sedation improves patient comfort and procedural efficiency, especially in complex cases, by reducing movement and coughing. However, it carries risks of respiratory depression and airway obstruction, potentially requiring premature termination or urgent intubation. Determining the optimal timing for intubation can be challenging despite proper monitoring. To enhance safety, the investigator has performed bronchoscopy under deep sedation with preemptive intubation for years, sharing this experience with other hospitals. This study aims to evaluate its safety and feasibility through a multicenter prospective observational approach.

DETAILED DESCRIPTION:
Bronchoscopy is a crucial procedure for diagnosing and treating respiratory diseases. It is recommended to be performed under sedation whenever possible, with sedation levels ranging from minimal to moderate and deep sedation. Deep sedation enhances patient comfort and facilitates the procedure, making it particularly useful for lengthy or complex bronchoscopic examinations. Additionally, deep sedation reduces involuntary patient movements and coughing, allowing the proceduralist to perform bronchoscopy more effectively when the patient is deeply sedated.

Despite its benefits, deep sedation carries the risk of respiratory depression and impaired airway maintenance, which may necessitate early termination of the bronchoscopy. If respiratory suppression or inadequate airway maintenance occurs during deep sedation, the procedure may need to be interrupted for endotracheal intubation using the bronchoscope. However, even with appropriate monitoring during bronchoscopy, determining the optimal timing for endotracheal intubation can be challenging, potentially disrupting procedural continuity and reducing the likelihood of a successful examination.

To enhance patient comfort and procedural safety, the investigator has been performing bronchoscopy under deep sedation with preemptive endotracheal intubation for several years. This clinical experience has been shared with other university hospitals in the region, and cases of deep sedation with preemptive intubation under the supervision of bronchoscopists have been reported. This study aims to evaluate the safety and feasibility of deep sedation with preemptive endotracheal intubation during bronchoscopy through a multicenter prospective observational approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a bronchoscopy-assisted procedure for diagnostic or therapeutic purposes
* Individuals who voluntarily consent to participate in the clinical study and sign a written informed consent form

Exclusion Criteria:

* Patients who have experienced acute myocardial infarction or acute stroke within the past six weeks
* Patients with contraindications to bronchoscopy (e.g., severe respiratory or cardiovascular comorbidities)
* Patients with a history of allergy to benzodiazepines, propofol, fentanyl, or flumazenil
* Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Patients with a severe hypersensitivity reaction to dextran 40
* Patients with a history of acute angle-closure glaucoma
* Pregnant women
* Prisoners
* Patients with psychiatric disorders
* Patients classified as ASA Physical Status IV or V by the American Society of Anesthesiologists (ASA)
* Any other patients deemed unsuitable for the clinical study by the investigator

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary lesions
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia during deep sedation under proceduralist guidance with endotracheal intubation | On the day of the bronchoscopy procedure, from the initiation of sedation therapy to the completion of the bronchoscopy procedure.
  This study investigates the incidence of hypoxia during deep sedation under the proceduralist's guidance with endotracheal intubation. Hypoxia is defined as an oxygen saturation of less than 94% sustained for more than 10 seconds during the procedure.

SECONDARY OUTCOMES:
The incidence of severe hypoxia during deep sedation under proceduralist guidance with endotracheal intubation | On the day of the bronchoscopy procedure, from the initiation of sedation therapy to the completion of the bronchoscopy procedure.
  This study investigates the incidence of hypoxia during deep sedation under the proceduralist's guidance with endotracheal intubation. Hypoxia is defined as an oxygen saturation of less than 90% sustained for more than 60 seconds during the procedure.
The incidence of complications | From the day of the bronchoscopy procedure to the outpatient visit one week after the procedure.
  early termination or delay of the procedure, complications from endotracheal intubation, complications from bronchoscopy
The rate of patient satisfaction | From the completion of the bronchoscopy procedure to the point when the patient has fully recovered from sedation.
  Patient satisfaction immediately after the procedure is assessed by two items: distress during fiberoptic bronchoscopy (distress/ tolerable/ no distress or satisfied) and willingness to be reexamined (accept/ never again).

CONTACTS AND LOCATIONS:
Overall Officials: Hee Yun Seol, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital, Yangsan, South Korea
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea